CLINICAL TRIAL: NCT03506555
Title: Laparoscopic Access in General Surgery: the Closed (Veress Needle) Technique Versus the Open (Hasson) Technique: A Randomised Controlled Trial
Brief Title: Laparoscopic Access in General Surgery: the Closed (Veress Needle) Technique Versus the Open (Hasson) Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sefako Makgatho Health Sciences University (Other)
Responsible Party: Principal Investigator, Dr Oleh Matsevych, Dr OY Matsevych (Department of Surgery), Sefako Makgatho Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: SefakoMSU
Record Dates: First submitted 2018-04-14; First posted 2018-04-24 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Laparoscopic Surgery; Laparoscopic Entry Technique
Keywords: Laparoscopy; Hasson technique; Veress needle technique; complications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the arm A (Veress needle) (Active Comparator): a standard reusable Veress needle technique was performed for laparoscopic entry
  Interventions: Procedure: Laparoscopic peritoneal entry technique: Veress needle versus Hasson
- the arm B (Hasson) (Active Comparator): the standard open Hasson technique was performed for laparoscopic entry
  Interventions: Procedure: Laparoscopic peritoneal entry technique: Veress needle versus Hasson

INTERVENTIONS:
Procedure: Laparoscopic peritoneal entry technique: Veress needle versus Hasson — According to randomization, the closed (Veress needle) or the open (Hasson) laparoscopic entry technique was utilized for general surgical operations

SUMMARY:
A randomised controlled trial (RCT) comparing the closed (Veress needle) with the open (Hasson) laparoscopic entry technique in haemodynamically stable patients undergoing either emergency or elective surgical procedures was conducted over a 13-month period. The success rate and complications related to the technique were recorded and analysed.

DETAILED DESCRIPTION:
A randomised controlled trial (RCT) was conducted at the single academic tertiary institution (Dr George Mukhari Academic Hospital (DGMAH), South Africa). Patients were recruited over a 13-month period (from 1st November 2014 to 30th November 2015). All haemodynamically stable patients undergoing either emergency or elective laparoscopic procedures were offered to participate in the study. General surgical patients 18 years or older who were eligible to provide an informed written consent were included in the study. Patients younger than 18 years old and haemodynamically unstable patients were excluded from the study. The success rate and complications related to the technique were recorded and analysed.

All included patients were randomised by computer program into one of two arms of the study: the arm A (Veress needle) or the arm B (Hasson). Participating surgeons were fully proficient with both techniques. The periumbilical area and the left hypochondrium (Palmer's point) were the recommended sites of entry, however, depending on clinical situation a surgeon could opt the other areas. In the A arm, a standard reusable Veress needle was used guided by tactile clicks feeling and water drop test. After pneumoperitoneum was established, the trocar was introduced in the same area. In the B arm, the standard open Hasson technique was used by dissecting tissues and dividing peritoneum between two forceps and introducing the port (a sleeve) without a trocar under direct visualization. Failed entry was defined as an inability to access the peritoneal cavity by a surgeon using the access technique initially selected.

An anonymized data collection form was completed by the general surgeon responsible for the procedure. Patients' age, gender, height, weight, diagnosis, type of surgery, previous abdominal surgery, previous abdominal tuberculosis (TB), primary port site placement, a surgeon, intraabdominal findings, complications and their type were recorded. Body Mass Index (BMI) was calculated and patients were categorised into weight groups: BMI above 30 and below 30.

All patients were followed up in 24 hours to detect the early entry-site complications. The complication after 24 hours, including surgical site infection and port-site hernia were not included in the design of this study.

ELIGIBILITY:
Inclusion Criteria:

* haemodynamically stable patients, undergoing either emergency or elective laparoscopic general surgical procedures

Exclusion Criteria:

* haemodynamically unstable patients, invalid consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2016-02-01 (Actual)

PRIMARY OUTCOMES:
the success rate | during surgery
  The technique resulted in establishment of pneumoperitoneum
complications/adverse events related to the technique | within 24 hours
  Any complications related to the technique

SECONDARY OUTCOMES:
Conditions leading to complications/adverse events | within 24 hours
  Any conditions leading to complications/adverse events were analyzed

IPD SHARING:
Plan to Share IPD: Undecided